CLINICAL TRIAL: NCT02734433
Title: A Phase 1 Study of Single Agent Pexidartinib in Asian Subjects With Advanced Solid Tumors
Brief Title: Study of Pexidartinib in Asian Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PL3397-A-A103
Record Dates: First submitted 2016-03-22; First posted 2016-04-12 (Estimated); Results first posted 2020-04-24 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-03

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced solid tumors; Asian subjects; Developmental Phase I
MeSH Terms: interventions — pexidartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: Yes

ARMS (1):
- Pexidartinib (Experimental): Pexidartinib capsules administered twice daily in the morning and evening. Each cycle of treatment is 28 days in duration. The cycle of treatment is continued until disease progression, unacceptable toxicity, or consent withdrawal.
  Interventions: Drug: Pexidartinib

INTERVENTIONS:
Drug: Pexidartinib

SUMMARY:
This is a Phase I, non-randomized, open-label, multiple dose study of pexidartinib in Asian subjects with advanced solid tumors. The study will be conducted in a dose escalation to assess the safety and tolerability, pharmacokinetics (PK) and pharmacodynamics (PD), and preliminary antitumor activity of pexidartinib.

ELIGIBILITY:
Inclusion Criteria:

* Age should be ≥ 20 years
* Subjects must have a pathologically documented solid tumor that has relapsed from, or is refractory to standard treatment, or for which no standard treatment is available
* All associated toxicity from previous cancer therapy must have been resolved (to ≤ Grade 1) prior to administration of pexidartinib
* Eastern Cooperative Oncology Group (ECOG) score of 0 or 1
* Adequate hematologic, hepatic, and renal function tests
* Adequate treatment washout period before registration defined as:

  1. Major surgery: ≥ 4 weeks (2 weeks for less invasive surgery, such as colostomy)
  2. Radiation therapy (eg, whole brain radiotherapy): ≥ 4 weeks (if palliative stereotactic radiation therapy, ≥ 2 weeks)
  3. Chemotherapy or immunotherapy (including targeted therapy with antibody or small molecule, retinoid therapy, and hormonal therapy): 4 weeks or 5 half-lives of the agent, whichever is shorter (if the regimen has contained nitrosoureas or mitomycin C, ≥ 6 weeks)
  4. Other investigational drug therapy: ≥ 4 weeks

Exclusion Criteria:

* Refractory nausea and vomiting, malabsorption, external biliary shunt, or significant small bowel resection that would have precluded adequate absorption
* Previous use of pexidartinib or any biologic treatment targeting colony stimulating factor-1 (CSF-1) or the receptor for colony-stimulating factor-1 (CSF1R); previous use of oral tyrosine kinase inhibitors, eg, imatinib or nilotinib, is allowed
* Clinically active primary central nervous system tumors or brain metastasis, defined as untreated and symptomatic, or requiring therapy with steroids or anticonvulsants to control associated symptoms
* Active or chronic infection with hepatitis C or known positive hepatitis B surface. antigen, or known active or chronic infection with human immunodeficiency virus
* A screening Fridericia-corrected time between the start of the Q wave and the end of the T wave in the heart's electrical cycle (QTcF) ≥ 450 ms (in men) or ≥ 470 ms (in women).
* A medical history or complications of clinically significant lung disease (eg, interstitial pneumonia, pneumonitis, pulmonary fibrosis, and severe radiation pneumonitis)
* A history of symptomatic congestive heart failure (CHF) [New York Heart Association (NYHA) Classes II to IV] or serious cardiac arrhythmia requiring treatment
* A history of myocardial infarction or unstable angina within 6 months before enrollment
* An uncontrolled infection requiring intravenous injection of antibiotics, antivirals, or antifungals

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-06-13 (Actual); Study Completion 2021-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (1):
- Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lewis JH, Gelderblom H, van de Sande M, Stacchiotti S, Healey JH, Tap WD, Wagner AJ, Pousa AL, Druta M, Lin CC, Baba HA, Choi Y, Wang Q, Shuster DE, Bauer S. Pexidartinib Long-Term Hepatic Safety Profile in Patients with Tenosynovial Giant Cell Tumors. Oncologist. 2021 May;26(5):e863-e873. doi: 10.1002/onco.13629. Epub 2020 Dec 24. PMID 33289960
- [Derived] Lee JH, Chen TW, Hsu CH, Yen YH, Yang JC, Cheng AL, Sasaki SI, Chiu LL, Sugihara M, Ishizuka T, Oguma T, Tajima N, Lin CC. A phase I study of pexidartinib, a colony-stimulating factor 1 receptor inhibitor, in Asian patients with advanced solid tumors. Invest New Drugs. 2020 Feb;38(1):99-110. doi: 10.1007/s10637-019-00745-z. Epub 2019 Mar 2. PMID 30825104

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 12 participants who met all inclusion and no exclusion criteria were enrolled in the study; 11 participants were treated.
Pre-assignment Details: The study was conducted in a dose-escalation 3 + 3 design and was comprised of 2 dose levels (Cohort 1 [600 mg/day] and Cohort 2 [1000 mg/day]). Selection of the pexidartinib dose of 1000 mg/day as the highest dose and the split-dose administration schedule was based on data from a Phase 1 study on patients with solid tumors (Study PLX108-01).
Groups:
- Cohort 1 - 600 mg/Day: Participants who received pexidartinib 600 mg/day (200 mg in the morning and 400 mg in the evening).
- Cohort 2 - 1000 mg/Day: Participants who received pexidartinib 1000 mg/day (400 mg in the morning and 600 mg in the evening) for the first 2 weeks. Thereafter, the dose was reduced to 800 mg/day (400 mg in the morning and 400 mg in the evening).
Period: Overall Study
Arm/Group | Cohort 1 - 600 mg/Day | Cohort 2 - 1000 mg/Day
Started | 3 | 8
Completed | 1 | 0
Not Completed | 2 | 8
Not completed — Disease progression | 1 | 5
Not completed — Clinical progression | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - 600 mg/Day | Cohort 2 - 1000 mg/Day | Total
Number analyzed (Participants) | 3 | 8 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 5 | 6
  >=65 years | 2 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (27.9) | 62.4 (12.2) | 60.4 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 2 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 8 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 3 | 8 | 11

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Based on RECIST V1.1 Following Oral Doses of Pexidartinib (Efficacy Analysis Set)
Description: For the assessment of tumor response, participants were classified into the best of the following tumor response categories by RECIST v1.1: complete response (CR), disappearance of all target lesions and normalization of tumor marker level; partial response (PR), at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters; stable disease (SD); neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study; progressive disease (PD), at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study and the sum must also demonstrate an absolute increase of at least 5 mm; or not evaluable (NE) for analysis. Objective response rate was defined as CR or PR and disease control rate was defined as CR, PR, or SD.
Time Frame: Day 1 through Day 28 after last dose (within 18 months)
Population: Best overall response was assessed in the Efficacy Analysis Set.
Measure: Number; unit: Number of participants
Arm/Group | Cohort 1 - 600 mg/Day | Cohort 2 - 1000 mg/Day
Number analyzed (Participants) | 3 | 5
Number of participants
  Complete response (CR) | 0 | 0
  Partial response (PR) | 1 | 0
  Stable disease (SD) | 1 | 3
  Progressive disease (PD) | 1 | 2
  Not evaluable (NE) | 0 | 0
  Objective response rate (CR or PR) | 1 | 0
  Disease control rate (CR or PR or SD) | 2 | 3

2. Secondary Outcome: Duration of Response or Duration of Stable Disease Following Oral Doses of Pexidartinib (Efficacy Analysis Set)
Description: Based on RECIST v1.1, complete response (CR), disappearance of all target lesions and normalization of tumor marker level; partial response (PR), at least a 30% decrease in sum of diameters of target lesions, with reference to baseline sum diameters; stable disease (SD); neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), with reference to smallest sum diameters; PD, at least a 20% increase in the sum of diameters of target lesions, with reference to smallest sum on study and sum must also demonstrate an absolute increase of at least 5 mm; Duration of response for responders (CR or PR) is defined as the time interval between the date of the earliest qualifying response and the date of PD or death for any cause, whichever occurs earlier. Duration of SD is defined as the time interval, in the absence of either CR or PR that will be calculated between the date of the first administration of the study drug and the date of PD.
Time Frame: Day 1 through Day 28 after last dose (within 18 months)
Population: Duration of response or duration of stable disease was assessed in the Efficacy Analysis Set.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Cohort 1 - 600 mg/Day | Cohort 2 - 1000 mg/Day
Number analyzed (Participants) | 1 | 3
months
  Duration of response (n=1,0): number analyzed (Participants) | 1 | 0
  Duration of response (n=1,0) | 7.62 (0) |
  Duration of stable disease (n=1,3) | 1.87 (0) | 4.62 (1.6)

3. Secondary Outcome: A Summary of Pexidartinib Pharmacokinetic Parameter (Cmax) by Cohort and Day Following Oral Doses of Pexidartinib
Description: Maximum concentration (Cmax) of pexidartinib was assessed using standard non-compartmental methods.
Time Frame: Cycle 1, Day 1 and Day 15 at predose, 0.5h, 1h, 2h, 4h, and 8h postdose (each cycle was 28 days)
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1 - 600 mg/Day | Cohort 2 - 1000 mg/Day
Number analyzed (Participants) | 3 | 8
ng/mL
  Day 1 | 3210 (1320) | 3650 (1170)
  Day 15: number analyzed (Participants) | 3 | 7
  Day 15 | 8490 (1430) | 10800 (2860)

4. Secondary Outcome: A Summary of Pexidartinib Pharmacokinetic Parameter (AUC[0-8h]) by Cohort and Day Following Oral Doses of Pexidartinib
Description: Area under the curve from 0 to 8 hours (AUC[0-8h]) was assessed using standard non-compartmental methods.
Time Frame: Cycle 1, Day 1 and Day 15 at predose, 0.5h, 1h, 2h, 4h, and 8h postdose (each cycle was 28 days)
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Cohort 1 - 600 mg/Day | Cohort 2 - 1000 mg/Day
Number analyzed (Participants) | 3 | 8
ng*h/mL
  Day 1 | 13300 (4720) | 16500 (4760)
  Day 15: number analyzed (Participants) | 3 | 7
  Day 15 | 50900 (18300) | 64600 (15900)

5. Secondary Outcome: A Summary of Pexidartinib Pharmacokinetic Parameter (Tmax) by Cohort and Day Following Oral Doses of Pexidartinib
Description: Time at maximum pexidartinib concentration (Tmax) was assessed using standard non-compartmental methods.
Time Frame: Cycle 1, Day 1 and Day 15 at predose, 0.5h, 1h, 2h, 4h, and 8h postdose (each cycle was 28 days)
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1 - 600 mg/Day | Cohort 2 - 1000 mg/Day
Number analyzed (Participants) | 3 | 8
hours
  Day 1 | 3.95 (3.51) | 2.48 (1.18)
  Day 15: number analyzed (Participants) | 3 | 7
  Day 15 | 1.00 (1.00) | 1.26 (0.94)

6. Secondary Outcome: A Summary of Pexidartinib Pharmacokinetic Parameter (R[AUC]) by Cohort Following Oral Doses of Pexidartinib
Description: Accumulation ratio of area under the curve (R[AUC]) was assessed using standard non-compartmental methods.
Time Frame: Cycle 1, Day 15 at predose, 0.5h, 1h, 2h, 4h, and 8h postdose (each cycle was 28 days)
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: accumulation ratio of AUC
Arm/Group | Cohort 1 - 600 mg/Day | Cohort 2 - 1000 mg/Day
Number analyzed (Participants) | 3 | 8
accumulation ratio of AUC | 4.29 (2.29) | 4.58 (2.23)

7. Secondary Outcome: A Summary of Pexidartinib Pharmacokinetic Parameter (R[Cmax]) by Cohort Following Oral Doses of Pexidartinib
Description: Accumulation ratio of maximum concentration of pexidartinib (R[Cmax]) was assessed using standard non-compartmental methods.
Time Frame: Cycle 1, Day 15 at predose, 0.5h, 1h, 2h, 4h, and 8h postdose (each cycle was 28 days)
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: accumulation ratio of Cmax
Arm/Group | Cohort 1 - 600 mg/Day | Cohort 2 - 1000 mg/Day
Number analyzed (Participants) | 3 | 8
accumulation ratio of Cmax | 2.94 (1.19) | 4.58 (2.23)

8. Secondary Outcome: A Summary of Plasma ZAAD-1006a Pharmacokinetic Parameter (AUC[0-8h]) Following Oral Doses of Pexidartinib
Description: Area under the curve from 0 to 8 hours (AUC[0-8h]) was assessed using standard non-compartmental methods.
Time Frame: Cycle 1, Day 1 and Day 15 at predose, 0.5h, 1h, 2h, 4h, and 8h postdose (each cycle was 28 days)
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Cohort 1 - 600 mg/Day | Cohort 2 - 1000 mg/Day
Number analyzed (Participants) | 3 | 8
ng*h/mL
  Day 1 | 14800 (8010) | 15600 (9130)
  Day 15: number analyzed (Participants) | 3 | 7
  Day 15 | 91600 (37500) | 120000 (61100)

9. Secondary Outcome: A Summary of Plasma ZAAD-1006a Pharmacokinetic Parameter (Cmax) Following Oral Doses of Pexidartinib
Description: Maximum concentration (Cmax) of pexidartinib was assessed using standard non-compartmental methods.
Time Frame: Cycle 1, Day 1 and Day 15 at predose, 0.5h, 1h, 2h, 4h, and 8h postdose (each cycle was 28 days)
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1 - 600 mg/Day | Cohort 2 - 1000 mg/Day
Number analyzed (Participants) | 3 | 8
ng/mL
  Day 1 | 2930 (935) | 3200 (1630)
  Day 15: number analyzed (Participants) | 3 | 7
  Day 15 | 13200 (5120) | 17800 (9630)

10. Secondary Outcome: A Summary of Plasma ZAAD-1006a Pharmacokinetic Parameter (Tmax) Following Oral Doses of Pexidartinib
Description: Time at maximum pexidartinib concentration (Tmax) was assessed using standard non-compartmental methods.
Time Frame: Cycle 1, Day 1 and Day 15 at predose, 0.5h, 1h, 2h, 4h, and 8h postdose (each cycle was 28 days)
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1 - 600 mg/Day | Cohort 2 - 1000 mg/Day
Number analyzed (Participants) | 3 | 8
hours
  Day 1 | 6.55 (2.24) | 5.00 (2.87)
  Day 15: number analyzed (Participants) | 3 | 7
  Day 15 | 1.5 (2.18) | 1.43 (0.87)

11. Secondary Outcome: A Summary of Plasma ZAAD-1006a Pharmacokinetic Parameter (MR AUC[0-8h]) Following Oral Doses of Pexidartinib
Description: Metabolite to parent drug ratio of area under the curve from 0-8 h (MR AUC[0-8h]) was assessed using standard non-compartmental methods.
Time Frame: Cycle 1, Day 1 and Day 15 at predose, 0.5h, 1h, 2h, 4h, and 8h postdose (each cycle was 28 days)
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: metabolite to parent drug ratio
Arm/Group | Cohort 1 - 600 mg/Day | Cohort 2 - 1000 mg/Day
Number analyzed (Participants) | 3 | 8
metabolite to parent drug ratio
  Day 1 | 0.801 (0.454) | 0.658 (0.298)
  Day 15: number analyzed (Participants) | 3 | 7
  Day 15 | 1.27 (0.416) | 1.33 (0.711)

12. Secondary Outcome: A Summary of Plasma ZAAD-1006a Pharmacokinetic Parameter (MR Cmax) Following Oral Doses of Pexidartinib
Description: Metabolite to parent drug ratio of maximum pexidartinib concentration (MR Cmax) was assessed using standard non-compartmental methods.
Time Frame: Cycle 1, Day 1 and Day 15 at predose, 0.5h, 1h, 2h, 4h, and 8h postdose (each cycle was 28 days)
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: metabolite to parent drug ratio
Arm/Group | Cohort 1 - 600 mg/Day | Cohort 2 - 1000 mg/Day
Number analyzed (Participants) | 3 | 8
metabolite to parent drug ratio
  Day 1 | 0.669 (0.189) | 0.639 (0.314)
  Day 15: number analyzed (Participants) | 3 | 7
  Day 15 | 1.10 (0.440) | 1.18 (0.695)

13. Secondary Outcome: Number and Percentage of Participants With Common Treatment-emergent Adverse Events (TEAEs) (≥20%) Classified by Preferred Term (Safety Analysis Set)
Description: An adverse event is any untoward medical occurrence in a subject administered a pharmaceutical product that does not necessarily have to have a causal relationship with this treatment. All TEAEs were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Event (NCI-CTCAE) Version 4.0.
Time Frame: Baseline through study completion, up to 18 months
Population: Adverse events were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - 600 mg/Day | Cohort 2 - 1000 mg/Day
Number analyzed (Participants) | 3 | 8
Participants
  Any TEAE | 3 | 8
  Chronic gastritis | 0 | 1
  Constipation | 0 | 2
  Diarrhoea | 0 | 3
  Nausea | 0 | 1
  Stomatitis | 0 | 1
  Face oedema | 0 | 1
  Fatigue | 1 | 3
  Malaise | 1 | 0
  Alanine aminotransferase increased | 1 | 3
  Aspartate aminotransferase increased | 2 | 3
  Blood alkaline phosphatase increased | 1 | 3
  Blood bilirubin increased | 1 | 1
  Blood cholesterol increased | 1 | 0
  Gamma-glutamyltransferase increased | 0 | 2
  Weight increased | 1 | 0
  Dysuria | 0 | 1
  Proteinuria | 1 | 0
  Urinary retention | 0 | 1
  Cough | 1 | 2
  Haemoptysis | 0 | 1
  Hair colour changes | 2 | 2
  Pruritus generalised | 1 | 0
  Rash generalised | 1 | 0
  Skin hypopigmentation | 0 | 1

14. Secondary Outcome: Number and Percentage of Participants With Treatment-related TEAEs by Preferred Term (Safety Analysis Set)
Description: as for outcome 13
Time Frame: Baseline through study completion, up to 18 months
Population: Adverse events were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - 600 mg/Day | Cohort 2 - 1000 mg/Day
Number analyzed (Participants) | 3 | 8
Participants
  Any treatment-related TEAE | 3 | 6
  Diarrhoea | 0 | 3
  Face oedema | 0 | 1
  Fatigue | 1 | 3
  Alanine aminotransferase increased | 1 | 3
  Aspartate aminotransferase increased | 2 | 3
  Blood alkaline phosphatase increased | 1 | 3
  Blood bilirubin increased | 1 | 0
  Blood cholesterol increased | 1 | 0
  Gamma-glutamyltransferase increased | 0 | 2
  Proteinuria | 1 | 0
  Hair colour changes | 2 | 2
  Pruritus generalised | 1 | 0
  Rash generalised | 1 | 0
  Skin hypopigmentation | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse event data were collected after the first dose up 28 days after the last dose through study completion, up to 18 months postdose.
Description: An adverse event is any untoward medical occurrence in a subject administered a pharmaceutical product that does not necessarily have to have a causal relationship with this treatment.
Arm/Group | Cohort 1 - 600 mg/Day | Cohort 2 - 1000 mg/Day
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/8
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/8
Other Adverse Events (participants affected / at risk) | 3/3 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 - 600 mg/Day (N=3) | Cohort 2 - 1000 mg/Day (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 - 600 mg/Day (N=3) | Cohort 2 - 1000 mg/Day (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Dacryostenosis acquired (Eye disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 3
Constipation (Gastrointestinal disorders) | 0 | 2
Chronic gastritis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 1 | 3
Face oedema (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 3
Alanine aminotransferase increased (Investigations) | 1 | 3
Blood alkaline phosphatase increased (Investigations) | 1 | 3
Blood bilirubin increased (Investigations) | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 2
Blood cholesterol increased (Investigations) | 1 | 0
Weight increased (Investigations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hair colour changes (Skin and subcutaneous tissue disorders) | 2 | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-25): https://cdn.clinicaltrials.gov/large-docs/33/NCT02734433/Prot_SAP_000.pdf